CLINICAL TRIAL: NCT06292091
Title: An Open-label, Fixed-sequence, 3-period Crossover Exploratory Study to Investigate the Effect of Urine Acid-base Disequilibrium on the Pharmacokinetics of Captopril in Healthy Male Volunteers
Brief Title: A Study to Investigate the Effect of Urine Acid-base Disequilibrium on the Pharmacokinetics of Captopril
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SeungHwan Lee, Associate Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Ur_ABD_PK
Record Dates: First submitted 2024-02-13; First posted 2024-03-04 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Captopril; Sodium Bicarbonate; Torsemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Captopril (Active Comparator): Single dose of captopril 12.5 mg
  Interventions: Drug: Captopril 12.5 Mg
- Sodium bicarbonate+captopril (Experimental): Single dose of captopril 12.5 mg during multiple doses of sodium bicarbonate 1 g every 4-6 hours
  Interventions: Drug: Captopril 12.5 Mg; Drug: Sodium bicarbonate 4 G
- Torsemide+captopril (Experimental): Single dose of captopril 12.5 mg during multiple doses of torsemide 20 mg every 6-12 hours
  Interventions: Drug: Captopril 12.5 Mg; Drug: Torsemide 20 MG

INTERVENTIONS:
Drug: Captopril 12.5 Mg — 12.5 mg of captopril
Drug: Sodium bicarbonate 4 G — 4 g of sodium bicarbonate
  Arms: Sodium bicarbonate+captopril
Drug: Torsemide 20 MG — 20 mg of torsemide
  Arms: Torsemide+captopril

SUMMARY:
The aim of this study is to evaluate the effect of urine acid-base disequilibrium on the pharmacokinetics of captopril in healthy male volunteers.

DETAILED DESCRIPTION:
* Pharmacokinetic analysis of captopril before and after urine acid-base imbalance
* Safety analysis

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer aged 19 to 50 years at screening
* Body weight between 50.0 kg and 90.0 kg and body mass index (BMI) between 18.5 kg/m2 and 29.9 kg/m2 at screening

  * Body Mass Index (kg/m2) = Weight (kg)/{Height (m)}2
* Participants who voluntarily decided to participate and agreed in writing to comply with study instructions after receiving sufficient explanation and complete understanding of the study
* Participants who are suitable as test subjects for this test as determined by the investigator through physical examination, clinical laboratory tests, and interviews, etc.

Exclusion Criteria:

* Participants who have or have a history of clinically significant hepatobiliary system (severe liver failure, viral hepatitis, etc.), kidney (severe renal impairment, etc.), nervous system, immune system, respiratory system, digestive system, endocrine system, blood/tumor, cardiovascular system (heart failure, Torsades de pointes, etc.), urinary system, mental system (mood disorder, obsessive-compulsive disorder, etc.), and sexual dysfunction, etc.
* Evidence or past history of gastrointestinal disease (Crohn's disease, gastrointestinal ulcer, gastritis, gastroesophageal reflux disease, etc.) or past history of gastrointestinal surgery (except for simple appendectomy and hernia repair) that might affect the safety and PK assessment of the investigational product.
* Hypersensitivity to drugs including captopril, sodium bicarbonate, and torsemide or other drugs (aspirin, antibiotics, etc.) or history of clinically significant hypersensitivity reactions
* Participants with genetic problems such as lactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Positive serum test (HBs antigen, HCV antibody, HIV antigen-antibody, and RPR) at screening
* Past history of alcohol and drug abuse or a positive urine test for drugs with abuse potential at screening
* Any abnormalities in vital signs after 3 minutes rest at screening

  * Systolic blood pressure < 90 mmHg or > 150 mmHg, Diastolic blood pressure < 60 mmHg or > 100 mHg
* QT/QTcF > 450 msec or any abnormalities on electrocardiogram (ECG) at screening
* Any abnormalities in blood tests at screening

  * AST (SGOT), ALT (SGPT) > 60 IU/L, creatinine clearance (CKD-EPI equation) < 80 mL/min
* Past or planned treatment with any prescription drugs or herbal medicine within 2 weeks, or any over the counter drugs, health functional foods, or vitamin supplements within 1 week, prior to the first scheduled dose (individual who is eligible based on other criteria may participate in the study at the discretion of the investigator).
* Participants who have taken drugs that induce drug-metabolizing enzymes such as barbiturates or inhibit drug metabolism such as clarithromycin within 1 month prior to the first scheduled dose
* Treatment with any investigational product in another clinical trial within 6 months prior to the first scheduled dose

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
AUClast of captopril | Pre-dose (0 hour) and up to 12 hours in each period
  Area under the concentration-time curve from 0 to last measurable concentration (AUClast)
Cmax of captopril | Observed value among pre-dose (0 hour) and up to 12 hours in each period
  Maximum concentration of captopril (Cmax)

SECONDARY OUTCOMES:
AUCinf of captopril | Pre-dose (0 hour) and up to 12 hours in each period
  Area under the concentration-time curve from 0 to infinite (AUCinf)
Tmax of captopril | Observed time point among pre-dose (0 hour) and up to 12 hours in each period
  Time to Cmax (Tmax)
t1/2 of captopril | Pre-dose (0 hour) and up to 12 hours in each period
  half-life (t1/2)
CL/F of captopril | Pre-dose (0 hour) and up to 12 hours in each period
  Apparent clearance (CL/F)
Vd/F of captopril | Pre-dose (0 hour) and up to 12 hours in each period
  Apparent volume of distribution (Vd/F)
fe of captopril | Pre-dose (0 hour) and up to 12 hours in each period
  Fraction of urinary excretion (fe)
urine pH | Pre-dose (0 hour) and up to 12 hours in each period
  urine pH
Safety parameters | Through study completion, an average of 3 months
  Number and frequency of participants observed adverse events in each period

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No